CLINICAL TRIAL: NCT00266617
Title: The Effect of Subcutaneous r-HuEPO in Patients With Chronic Anemia Secondary to Chemotherapy
Brief Title: A Study to Evaluate the Safety and Effectiveness of Epoetin Alfa in Patients With Anemia as a Result of Advanced Cancer and Treatment With Aggressive Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005845
Record Dates: First submitted 2005-12-16; First posted 2005-12-19 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Neoplasms
Keywords: Anemia; chemotherapy; epoetin alfa; epogen; erythropoietin; neoplasms; cancer
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of epoetin alfa in the treatment of persistent anemia caused by advanced cancer and aggressive adriamycin-chemotherapy. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Patients undergoing treatment with adriamycin-containing chemotherapy frequently develop significant anemia. Agents that can increase the amount of hemoglobin in cancer patients undergoing treatment with non-platinum-containing cyclic chemotherapy may improve the patients' reduced physical strength and reduced stamina resulting from anemia, improve the patients' ability to continue chemotherapy, and improve the patients' overall qualify of life. Epoetin alfa is a genetically engineered form of a natural hormone, erythropoietin, that is used to treat anemia by stimulating red blood cell production. This is a randomized, double-blind, placebo-controlled, parallel group, multicenter study. The study evaluates the safety and effectiveness of epoetin alfa in treating patients who develop persistent anemia as a result of treatment with aggressive non-platinum-containing cyclic chemotherapy for any cancer type (except rapid and severe onset of leukemias and malignancies of the bone marrow and spleen). The study consists of a screening period when patients' eligibility is determined, a 12-week double-blind treatment period when patients receive 3 injections each week with either epoetin alfa or placebo, and an optional open-label treatment period when patients who choose to continue will receive 3 injections of epoetin alfa per week during any remaining cycles of their chemotherapy. Eligible patients will be randomly assigned to one of two treatment groups: one group receiving epoetin alfa 150 units/kilogram and the other group receiving a comparable volume of placebo. Study drug is administered by injection beneath the skin 3 times weekly for 12 weeks. The dose of study medication may be increased or decreased at the discretion of the physician, based on the results of blood tests. Depending on the patient's chemotherapy cycle, he or she will return to the study site every 3 or 4 weeks for administration of study medication. Safety evaluations (laboratory tests, vital sign measurements, reporting of adverse events, physical examination, and electrocardiogram) are performed throughout the study. The primary measures of effectiveness of the study drug will be determined by the number of transfusions patients require and by changes in blood test results for hemoglobin, hematocrit, and reticulocytes (immature red blood cells) from before the start of the study to the end of the study. The study hypothesis is that epoetin alfa will, more effectively than placebo, stimulate adequate production of red blood cells to increase the hemoglobin level in cancer patients who are anemic as a result of undergoing treatment with aggressive non-platinum-containing cyclic chemotherapy. Double-blind: Epoetin alfa 150 units/kilogram (U/kg) or matching volume placebo injected beneath the skin 3 times weekly for 12 weeks. Open-label: Epoetin alfa at the dose received at the end of the double-blind study injected beneath the skin 3 times weekly for any remaining cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer (except for rapid onset of severe leukemia and malignancies of the bone marrow and spleen) and anemia resulting from non-cisplatin-containing chemotherapy who are receiving cyclic chemotherapy for <=5 consecutive days every 3 or 4 weeks (for 3 cycles of chemotherapy)
* having a Performance score of 0, 1, 2, or 3 (patients' ability to perform daily activities, a self-care performance score of 0 [fully active, no disease restriction] to 3 [capable of only limited self-care, confined to bed or chair more than 50% of waking hours])
* having a life expectancy of at least 3 months
* with signs and symptoms of physical stability for 1 month before the study, (based on physical examination including vital signs, weight, and electrocardiogram), not grossly obese, and having a hemoglobin <= 10.5 grams/deciliter (g/dL)
* who are able to demonstrate the ability to administer self-injections

Exclusion Criteria:

* Patients with a history of any blood disease
* having signs and symptoms of significant disease/dysfunction not caused by the underlying cancer
* having a spread of cancer to the brain
* having uncontrolled high blood pressure, an iron, folate or vitamin B12 deficiency, or a history of seizures
* received therapy with androgen within 2 months before the start of study, received radiation therapy or surgery to decrease the number of cancer cells within 30 days before the start of the study, or experienced sudden and severe onset of illness within 7 days before the start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Study Completion 1990-06 (Actual)

PRIMARY OUTCOMES:
Number of transfusions; Change from baseline in levels of hemoglobin, hematocrit, reticulocytes (immature red blood cells)

SECONDARY OUTCOMES:
Change from baseline to end of study in: Quality of life; Physician's Global Evaluation of Study Medication; Patient's performance scores (energy level and daily activities); Assessment of safety

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study to evaluate the safety and effectiveness of epoetin alfa given by injection beneath the skin to patients with anemia as a result of advanced cancer and treatment with aggressive chemotherapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=674&filename=CR005845_CSR.pdf